CLINICAL TRIAL: NCT04503681
Title: A Pre-consultation Compassion Intervention to Reduce Anxiety Among Patients Referred to a Cancer Center
Brief Title: Pre-consultation Compassion Among Patients Referred to a Cancer Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Brian Roberts, Study Director, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-009
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Anxiety; Compassion; Empathy
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard introduction video (Active Comparator)
  Interventions: Other: Standard introduction video
- Enhanced compassion video (Experimental)
  Interventions: Other: Enhanced compassion video

INTERVENTIONS:
Other: Enhanced compassion video — Added five additional sentences to the standard introduction video. Those five sentences were compassion-focused statements. The compassionate statements added to the "enhanced compassion video" were based on the results of a recent systematic review of clinician compassionate behaviors, which found incorporating statements of support, acknowledgement, patient's perspective, emotion naming, and validation increased patient perception of compassion.
  Arms: Enhanced compassion video
Other: Standard introduction video — Standard introduction video sent to a new patient via email introducing the new patient to the cancer center prior to the initial consultation.
  Arms: Standard introduction video

SUMMARY:
Patients diagnosed with cancer commonly have a high degree of anxiety during an initial oncology consultation, which may interfere with a patient's ability to retain information required to make informed treatment decisions. A previous study randomized breast cancer survivors (volunteers) to view either (a) a brief video depicting a standard initial consultation from an oncologist or (b) an identical consultation with the addition of compassionate statements from the oncologist, and found the compassionate statements reduced anxiety among the volunteers. However, it is currently unknown if watching a video containing compassionate statements from an oncologist prior to an actual initial oncology consultation will reduce anxiety among patients referred to a cancer center. The aim of this randomized control trial is to test if watching a brief video containing compassionate statements from an oncologist, compared to watching a standard introduction video, prior to an initial oncology consultation will reduce the degree of anxiety among patients referred to a cancer center.

This is a prospective, randomized controlled clinical trial at an academic cancer center. The investigators will enroll adult patients scheduled for an initial oncology consultation. Subjects will be randomly assigned to receive a "standard introduction video" or "enhanced compassion video" for viewing prior to the initial oncology consultation. On arrival to the cancer center anxiety severity will be measured using the Hospital Anxiety and Depression scale (HADS). The HADS has two 7-item subscales (HADS Anxiety and HADS Depression) and is well-validated among oncology patients. Wilcoxon rank-sum test will be used to test for a difference in the HADS subscales between the two video groups.

DETAILED DESCRIPTION:
Study design This study is a prospective, randomized, controlled, parallel-group clinical trial at a single university-based cancer center (MD Anderson Cancer Center at Cooper, Cooper University Health Care, Camden, New Jersey, USA). Potential subjects will be enrolled at the time of scheduling an initial cancer consultation. The Cooper University Hospital Institutional Review Board allowed alteration of the requirements of obtaining informed consent under 45 CFR 46.116(d) given the intervention was deemed no greater than minimal risk. All new adult patients scheduled for an initial cancer consultation at MD Anderson Cancer Center at Cooper will be randomized to receive an email containing a link for either the "standard introduction video" or the "enhanced compassion video." Emails will be sent to patients prior to obtaining informed consent to allow for viewing of the video prior to the initial oncology consultation and to keep the patients masked to the study hypotheses prior to the consultation. When the patients arrive to the MD Anderson Cancer Center waiting room for his/her initial cancer consultation they will be approached by research staff to obtain written informed consent to complete the research questionnaire and for use of data.

Randomization and masking Patients will be randomly assigned to one of two groups, "standard introduction video" or "enhanced compassion video." An independent statistician will generate the group assignment sequence using a parallel design, 1:1 randomization schedule. Standard measures will be used to ensure appropriate concealment of group assignment. The randomization assignments will be kept in a sequential list and maintained in the scheduling operator office. At the time of scheduling an initial consultation, appointment operators will identify the next assignment in the series, which will be labeled either "Video A" or "Video B." The operators will then send the appropriate email containing a link to a website for the matching video. The independent statistician will maintain the code link for the videos. Thus, the operators, investigators, and research statistician will be blinded to video allocation until after all study analyses have been completed.

Interventions As part of a currently ongoing clinical quality initiative at the study institution, when a new patient schedules an appointment for an initial cancer consultation the scheduling operator sends an email to the patient containing a link for a standard introduction video. For the purposes of this study a second "enhanced compassion video" was developed, which added five additional sentences to the standard introduction video. Those five sentences were compassion-focused statements. Both videos feature the same oncologist (i.e. Medical Director of MD Anderson Cancer Center at Cooper) and are identical aside from the additional compassionate statements. The compassionate statements added to the "enhanced compassion video" were based on the results of a recent systematic review of clinician compassionate behaviors, which found incorporating statements of support, acknowledgement, patient's perspective, emotion naming, and validation increased patient perception of compassion.

Measurements and Data Collection After obtaining written informed consent a research questionnaire will be administered to patients at the cancer center prior to the initial cancer consultation. The questionnaire will assess the patients' perception of the video oncologist's compassion using the 5-item compassion measure, a previously validated patient-assessed measure of perceived compassion during patient care. Subject demographics, as well as clinical information pertaining to cancer diagnosis will be abstracted from the medical record.

Outcome measures The primary outcome measure will be anxiety severity on arrival to the cancer center for the initial consultation. As part of the research questionnaire subjects will be asked to complete the Hospital Anxiety and Depression scale (HADS). The HADS is a 14-item self-reported instrument that assesses anxiety and depressive symptoms in populations with medical conditions (both in- and out-patients). It has two 7-item subscales: HADS Anxiety and HADS Depression. Each item is scored on a 4-point scale (0=not at all to 3=nearly all the time); thus, each sub-scale can range from 0-21. The HADS has been extensively validated in oncology populations, and is a commonly used measure of anxiety and depression in oncology studies. The HADS Depression score will be analyzed as a secondary outcome. An additional secondary outcome measure will be the no-show rate for the initial consultation among each group. All data will be entered into Research Electronic Data Capture (REDCap), a secure, web-based application designed to support data capture for research studies, and export the data into Stata/SE 16.0 for Mac, StataCorp LP (College Station, TX, USA) for analysis.

Statistical analysis For descriptive statistics categorical data will be reported as proportions with 95% confidence intervals and continuous data as means with standard deviations or medians with interquartile ranges as appropriate. As part of the CONSORT diagram the proportion of patients who do not attend their initial cancer consultation, as well as the proportion of patients who attend their initial consultation, but decline to participate in the study, will be recored and stratified by video group. The investigators will test if the "enhanced compassion video" reduced the no-show rate to the initial consultation, as well as increased participation in research using the Fisher exact test. Cronbach's alpha will be used to separately test the internal reliability of the HADS anxiety scale, HADS depression scale, and the 5-item compassion measure among our cohort. The investigators will test if the "enhanced compassion video" group perceived the video oncologist as more (or less) compassionate, as measured by the 5-item compassion measure, than the "standard introduction video" group using the Wilcoxon rank-sum test.

For the primary outcome, the Wilcoxon rank-sum test will be used to test for a difference in the HADS anxiety scale between the two video groups. Sensitivity analysis dichotomizing the HADS anxiety scale into low (< 8) and moderate/high (≥ 8) will be performed. A cut point of 8 on the HADS subscales has been defined as the optimal cut point for diagnosis screening and is commonly used to define clinically significant symptoms in research studies. The Fisher exact test will be used to test if the proportion of subjects with clinically significant symptoms differed between the two video groups. For the secondary outcome measure the investigators will repeat the same analyses described above using the HADS depression scale in place of the HADS anxiety scale. The investigators will perform the above analyses using intention to treat methodology. The analyses will be repeated in a per protocol fashion excluding patients who state they did not watch the video prior to presentation to the cancer center.

To test if the relationship between video group and anxiety severity differs among pre-specified subgroups the investigators will perform separate multivariable linear regression models with the HADS anxiety scale as the dependent variable, and entering the following patient characteristic along with an interaction term between video group and the characteristic as independent variables: (1) age (decile), (2) sex (male vs. female), (3) race (white vs. non-white), (4) ethnicity (Hispanic vs. non-Hispanic), (5) suspected primary cancer (breast vs. gastrointestinal vs. pulmonary vs. skin vs. central nervous system vs. gynecologic vs. other).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* scheduled for an initial oncology consultation

Exclusion Criteria:

* patients who do not have an active email address or are medically unable to complete the research questionnaire at the time of the initial cancer consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
After review and approval by our study data use committee, we will allow other researchers who submit to us a suitable protocol to have access to the complete de-identified datasets used and/or analyzed during the study, in comma separated value format together with a data dictionary.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Winn C, Grana G, Mazzarelli A, Nicholson A, Mykulowycz K, Obiakor C, Bair A, Trzeciak S, Roberts B. Preconsultation compassion video to reduce anxiety among patients referred to a cancer centre: a randomised control trial. BMJ Oncol. 2024 Aug 6;3(1):e000427. doi: 10.1136/bmjonc-2024-000427. eCollection 2024. PMID 39886127
- [Derived] Winn C, Generosa G, Mazzarelli A, Trzeciak S, Roberts BW. Preconsultation compassion intervention to reduce anxiety among patients referred to a cancer center: protocol for a randomised control trial. BMJ Open. 2021 May 24;11(5):e048201. doi: 10.1136/bmjopen-2020-048201. PMID 34031118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Introduction Video | Enhanced Compassion Video
Started | 188 | 186
Completed | 183 | 179
Not Completed | 5 | 7
Not completed — Subjects did not complete outcome questionnaire | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Introduction Video | Enhanced Compassion Video | Total
Number analyzed (Participants) | 188 | 186 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13) | 62 (11) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 117 | 238
  Male | 67 | 69 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 179 | 179 | 358
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 26 | 54
  White | 129 | 133 | 262
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS)
Description: Seven item subscale. Each item is scored on a 4-point scale (0=not at all to 3=nearly all the time); thus, range from 0-21. Higher score indicates greater anxiety.
Time Frame: Baseline (on arrival to the cancer center for an initial oncology consultant).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Introduction Video | Enhanced Compassion Video
Number analyzed (Participants) | 183 | 179
score on a scale | 7 [4 to 10] | 7 [4 to 10]
Statistical Analysis 1: Comparison: Standard Introduction Video vs Enhanced Compassion Video; Test type: Superiority; p = 0.473, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1.1 to 1.1]

2. Secondary Outcome: Depression Subscale of the Hospital Anxiety and Depression Scale
Description: Seven item subscale. Each item is scored on a 4-point scale (0=not at all to 3=nearly all the time); thus, range from 0-21. Higher score indicates greater depression
Time Frame: Baseline (on arrival to the cancer center for an initial oncology consultant).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Introduction Video | Enhanced Compassion Video
Number analyzed (Participants) | 183 | 179
score on a scale | 3 [1 to 6] | 3 [1 to 6]
Statistical Analysis 1: Comparison: Standard Introduction Video vs Enhanced Compassion Video; Test type: Superiority; p = 0.338, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.8 to 0.8]

ADVERSE EVENTS:
Time Frame: At the time of oncology consultation and administration of the research questionnaire. Median (interquartile range) 9 (5 - 15) days after the introduction videos were emailed.
Arm/Group | Standard Introduction Video | Enhanced Compassion Video
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/186
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/186
Other Adverse Events (participants affected / at risk) | 0/188 | 0/186

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04503681/Prot_SAP_000.pdf